CLINICAL TRIAL: NCT04662346
Title: Difficulty Scoring System in Robotic Pancreatoduodenectomy
Brief Title: Evaluation of Difficulty Score for Robotic Pancreatoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Concetta Cacace, principal investigator, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Difficulty Score RPD
Record Dates: First submitted 2020-11-30; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients undergoing robotic pancreatoduodenectomy (Other): patients have pancreatic neoplasm and undergoing robotic pancreatoduodenectomy
  Interventions: Other: Difficulty score system for robotic pancreatoduodenectomy

INTERVENTIONS:
Other: Difficulty score system for robotic pancreatoduodenectomy — calculate the score for patient in you cohort

SUMMARY:
Robotic pancreatoduodenectomy is the most complex surgery for a general surgeon and consequently a pancreatic surgeon can aspire to. Due to the close proximity of the pancreas to the large vessels, great skill and experience in the field of pancreatic surgery, robotic surgery and also vascular surgery is essential. The ability to predict the depth of robotic pancreatoduodenectomy in each individual patient would be extremely important, for patient selection and for the implementation of the learning curve. This study aims to provide a difficulty score (DS) for robotic pancreatoduodenectomy to be used to select cases based on the experience and expertise of the surgeon.

DETAILED DESCRIPTION:
Our Robot DIFFICULT Score was developed starting from factors evaluated by surgeons with experience in performing robotic pancreatoduodenectomy in high-volume centers. Based on the univariate and multivariate analysis, the elevated BMI, ASA 3, the need for venous resection and vascular variations in arterial liver supply were considered significant in increasing the degree of "difficulty" in the robotic pancreatoduodenectomy. The Robot ADDICT Score will be calculated in all cases of the International Consortium on Minimally Invasive Pancreatic Surgery (I-MIPS; www.i-mips.com).

ELIGIBILITY:
Inclusion Criteria:

* pathology of the head of pancreas requiring surgery

Exclusion Criteria:

* pathology of the head of pancreas not requiring surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
correlation to post-operative complication | 6 months
  the score increase as complications increase

CONTACTS AND LOCATIONS:
Overall Officials: ugo boggi, Study Chair — University of Pisa
Locations (2):
- Italy (2):
  - Division of pancreatic surgery, Pisa
  - University of Pisa, Pisa

IPD SHARING:
Plan to Share IPD: Yes
creation of the formula, validation
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 month
Access Criteria: surgeon

REFERENCES:
- [Derived] Napoli N, Cacace C, Kauffmann EF, Jones L, Ginesini M, Gianfaldoni C, Salamone A, Asta F, Ripolli A, Di Dato A, Busch OR, Cappelle ML, Chao YJ, de Wilde RF, Hackert T, Jang JY, Koerkamp BG, Kwon W, Lips D, Luyer MDP, Nickel F, Saint-Marc O, Shan YS, Shen B, Vistoli F, Besselink MG, Hilal MA, Boggi U; International Consortium on Minimally Invasive Pancreatic Surgery (I-MIPS). The PD-ROBOSCORE: A difficulty score for robotic pancreatoduodenectomy. Surgery. 2023 Jun;173(6):1438-1446. doi: 10.1016/j.surg.2023.02.020. Epub 2023 Mar 25. PMID 36973127